CLINICAL TRIAL: NCT04813692
Title: Mechanical Complications of Acute Myocardial Infarction: an International Multicenter Cohort Study During COVID-19 Pandemics (CautionCov19)
Brief Title: Mechanical Complications of Acute Myocardial Infarction During COVID-19 Pandemics
Acronym: CautionCov19
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IT-VA:85/2021
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Ventricular Septal Rupture; Papillary Muscle Rupture; Free Wall Rupture, Heart
MeSH Terms: conditions — Ventricular Septal Rupture; Heart Rupture | interventions — Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical repair — Surgical repair of post-infarction LVFWR or VSR
Procedure: Percutaneous treatment — Percutaneous closure of post-infarction VSR (or treatment for LVFWR)
Procedure: Mitral valve surgery — Mitral valve repair or replacement for post-infarction PMR

SUMMARY:
The ongoing COVID-19 pandemics has put an overwhelming pressure on the healthcare systems of many European countries. Such a situation has potentially led to delayed and impaired access to appropriate treatment for patients affected by other severe, non-COVID-19-related conditions, including cardiovascular diseases. This resulted in a reported lower admission, but higher mortality rate for AMI patients.

Such a situation might be explained by many factors, including unavailability of early reperfusion therapy and late hospital presentation of AMI patients due to a general anxiety related to the COVID-19 contagious risk of the hospital environment. As a matter of fact, during this year of pandemics, several case reports suggested a new, significant surge of post-AMI mechanical complications, sometimes describing patients admitted in too severe conditions to consider surgical repair a viable option, and therefore inevitably undergone an unfavorable outcome.

Therefore, we decided to involve the large network of European centers already participating to the "Caution Study 1", in order to study the impact of COVID-19 pandemics on the outcomes, incidence and treatments of post-AMI mechanical complications.

DETAILED DESCRIPTION:
Mechanical complications must be carefully searched for in any patient with an acute coronary syndrome and signs of cardiogenic shock, as prompt diagnosis and immediate surgery often represent the only effective treatment for such ominous conditions.

The management of patients with postinfarction mechanical complications requires the consideration of several factors: (i) the extremely poor prognosis without surgical treatment; (ii) the higher mortality risk associated with emergency surgery; (iii) the potential rapid deterioration of initially stable patients.

Data from the Society of Thoracic Surgeons National Database demonstrated an average 43% in-hospital/30-day mortality for surgical treatment of ventricular septal rupture. Data from the same registry on papillary muscle rupture showed a 30-day mortality of 20%. Matteucci et al. recently reported a 36.4% mortality rate for free wall rupture from the large CAUTION multicenter study.

Given the low incidence of these post-AMI mechanical complications, evidence-based therapeutic strategies remain controversial, and little is known on the early clinical results and late follow-up, with most information derived from small single-center experiences or national registries.

Therefore, we started the "Mechanical complications of acute myocardial infarction: an international multicenter cohort study" - (Caution Study 1), a retrospective, international multicenter clinical trial aimed at evaluating the survival, postoperative outcome and quality of life of patients undergone cardiac surgery for post-infarction mechanical complications starting from 2001.

The ongoing COVID-19 pandemics, however, has put an overwhelming pressure on the healthcare systems of many European countries. Such a situation has potentially led to delayed and impaired access to appropriate treatment for patients affected by other severe, non-COVID-19-related conditions, including cardiovascular diseases. This resulted in a reported lower admission, but higher mortality rate for AMI patients.This situation might be explained by many factors, including unavailability of early reperfusion therapy and late hospital presentation of AMI patients due to a general anxiety related to the COVID-19 contagious risk of the hospital environment. As a matter of fact, during this year of pandemics, several case reports suggested a new, significant surge of post-AMI mechanical complications, sometimes describing patients admitted in too severe conditions to consider surgical repair a viable option, and therefore inevitably undergone an unfavorable outcome.

Therefore, we decided to involve the large network of European centers already participating to the "Caution Study 1", in order to study the impact of COVID-19 pandemics on the outcomes, incidence and treatments of post-AMI mechanical complications.

"Mechanical complications of acute myocardial infarction: an international multicenter cohort study during COVID-19 pandemics" is a retrospective, international multicenter clinical trial aimed at evaluating the trend of incidence, types of treatment and survival of patients admitted to hospital with a diagnosis of post-infarction mechanical complications.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old;
* recent diagnosis of acute myocardial infarction;
* presence of ventricular free-wall rupture and/or ventricular septal rupture and/or papillary muscle rupture.

Exclusion Criteria:

* patients < 18 years old;
* ventricular free-wall rupture or ventricular septal rupture or papillary muscle rupture not related with acute myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who were diagnosed with mechanical complications of acute myocardial infarction, between March 2018 to February 2021, independent of the treatment offered.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
In-hospital survival | interval from intervention (surgical or percutaneous) to hospital discharge (expected: up to 4 weeks)
  To assess the in-hospital survival rate of patients admitted with a diagnosis of post-AMI mechanical complications and underwent surgical or percutaneous treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Matteucci Matteo, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided